CLINICAL TRIAL: NCT02823691
Title: Safety of Lanreotide 120 mg ATG in Combination With Metformin in Patients With Progressive Advanced Well-differentiated Gastro-intestinal (GI) or Lung Carcinoids: A Pilot, One-arm, Open-label, Prospective Study: the MetNET-2 Trial
Brief Title: The MetNET-2 Trial
Acronym: MetNET-2
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Cecilia Melani, MD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NationalCIMilan
Record Dates: First submitted 2016-05-19; First posted 2016-07-06 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Neuroendocrine Tumors
Keywords: NETs
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lanreotide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lanreotide and Metformin (Experimental): Dose and Treatment Regimen:
  LANREOTIDE ATG 120 mg/28 days (equivalent to 1 cycle), deep subcutaneous injection (SC) in combination with METFORMIN 2550 mg daily (maximum dose), oral administration (OS).
  Metformin starting dose 850 mg/day to be increased up to 1700 mg/day at day 14, 2550 mg/day at day 28, (maximum dose), if well tolerated.
  Interventions: Drug: Lanreotide and Metformin

INTERVENTIONS:
Drug: Lanreotide and Metformin — Lanreotide and Metformin
  Other Names: Ipstyl and Metformin

SUMMARY:
This is a Pilot, One-arm, Open-label, Prospective Study to evaluate Safety of Lanreotide 120 mg ATG in combination with Metformin in patients with advanced progressive GI or lung carcinoids.

The patient population will include patients with a histologically documented diagnosis of Well differentiated NET, G1-G2 according to the last WHO Classification criteria for GI and lung NET carcinoids.

DETAILED DESCRIPTION:
This study is strategically positioned in the medical treatment safety and efficacy context, that is Lanreotide can be safely and effectively used in combination with other agents, like Metformin.

Aim of this study is to verify the safety of a concomitant administration of Lanreotide 120 mg ATG with Metformin in advanced, progressing gastro-intestinal or lung carcinoids patients, by accurately monitor patients from a tolerability point of view during all study long.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (male or female, age > 18 years)
* Patient with advanced disease, not resectable. The evaluation of unresectable disease will be performed by surgeon of multidisciplinary Milan ENETS Center of Excellence tumour board of Fondazione IRCCS Istituto Nazionale dei Tumori Milano.
* Patients with a histologically documented diagnosis of advanced well differentiated (G1 and G2) GI or lung carcinoids, defined according to the last WHO Classification criteria for NET
* Tumor tissue available for analysis
* Measurable disease and disease progression in the 6 months before study inclusion (according to RECIST vs 1.1), documented and appropriate imaging
* Patient who has received prior treatment with surgery or chemotherapy or somatostatin analogues or m-TOR inhibitors or other systemic antineoplastic/target therapies
* Functioning or non-functioning NETs
* Type-2 Diabetic or normoglycaemic patient
* Documented Octreoscan/PET Ga68 uptake/IHC stain of SSTR2 receptor, within 6 months before study entry
* Basal blood tests:
* Counts of neutrophils in absolute value> 1.5 x 103 / L
* Platelet count> 100 x 103 / L
* Hemoglobin> 9 g/dl
* Total Bilirubin <1.5 times the upper limit of normal
* AST, ALT <2.5 times the upper limit of normal
* Alkaline phosphatase <2.5 times the upper limit of normal
* Values of serum creatinine <1.5 mg / dl. - CCr ≥ 60 mL / min
* ECOG performance status ≤ 2
* Life expectancy > 12 months
* Written informed consent
* Female subjects of childbearing potential (not surgically sterile or 2 years postmenopausal) must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for at least 60 days after participation in the study. Acceptable methods of contraception include double barrier method [i.e. condom and occlusive cap (diaphragm or cervical/vault caps)] spermicide, intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.
* Male subjects with female partners of childbearing potential must use a medically accepted method of contraception and must agree to continue use of this method for the duration of the study and for 60 days after participation in the study.

Exclusion Criteria

* Surgery performed within 28 days prior to the beginning of study treatment
* Brain metastasis or spinal cord compression
* Type-1 Diabetes
* Clinically significant cardiovascular disease, such as cardiovascular accidents occurred in less than 6 months, unstable angina, congestive heart failure grade greater than or equal to II (according to the classification of the New York Heart Association NYHA) series cardiac arrhythmias that require treatment
* Uncontrolled high blood pressure, atrial fibrillation
* Cardio-vascular, lung, kidney or hepatic disorders not treated/controlled
* Cirrhosis, acute hepatitis or chronic active hepatitis
* Metabolic disorders, clinical examination or laboratory investigations which contraindicate the use of drugs to study, or patients at high risk of complications from the treatment
* Active or uncontrolled severe infections
* Patients with a condition of metabolic acidosis, acute or chronic, including ketoacitosi
* History of POTUS (alcohol abuse), or habitual intake of alcohol (≥ 3 glasses of alcoholic drinks / day) sufficient to cause hepatotoxicity
* Severe states of dehydration
* Prolonged fasting
* History of immunosuppression, including positive HIV test
* Previous or concomitant oncological pathology, except: basal cell skin cancer, in situ, as long as every other cancer patient disease-free for at least 5 years
* Serious neurological or psychiatric disorders
* Pregnancy or lactation
* Patients that do not use appropriate methods of contraception as specified in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
incidence of SAEs and AEs | 1 year

SECONDARY OUTCOMES:
time to progression (TTP) to Lanreotide ATG 120 mg in combination with Metformin | 3 years
  This is a pilot study. This endpoints should be considered an exploratory evaluation
symptomatic responses to Lanreotide ATG 120 mg in combination with Metformin in symptomatic patients | 1 year
  Answers will be based on a 5 point Likert scale (1=completely satisfied, 2= rather satisfied, 3= unchanged, 4= rather dissatisfied, 5= completely dissatisfied).
biochemical responses to Lanreotide ATG 120 mg in combination with Metformin | 1 year
  Biochemical progression will be evaluated testing Chromogranin A, NSE, 5-HIAA (only if functioning tumours) at each 4th month

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pusceddu, MD, Principal Investigator
Locations (1):
- NationalCIMilan, Milan, Italy

REFERENCES:
- [Background] Culler MD, Oberg K, Arnold R, Krenning EP, Sevilla I, Diaz JA. Somatostatin analogs for the treatment of neuroendocrine tumors. Cancer Metastasis Rev. 2011 Mar;30 Suppl 1:9-17. doi: 10.1007/s10555-011-9293-0. PMID 21369878
- [Background] Rizos CV, Elisaf MS. Metformin and cancer. Eur J Pharmacol. 2013 Apr 5;705(1-3):96-108. doi: 10.1016/j.ejphar.2013.02.038. Epub 2013 Mar 13. PMID 23499688
- [Background] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687
- [Background] Vlotides G et Al: anticancer effects of metformin on neuroendocrine tumor cell in vitro. 10 the ENETs Annual conference Barcelona 5-8 March 2013
- [Background] Evans JM, Donnelly LA, Emslie-Smith AM, Alessi DR, Morris AD. Metformin and reduced risk of cancer in diabetic patients. BMJ. 2005 Jun 4;330(7503):1304-5. doi: 10.1136/bmj.38415.708634.F7. Epub 2005 Apr 22. No abstract available. PMID 15849206
- [Background] Decensi A, Puntoni M, Goodwin P, Cazzaniga M, Gennari A, Bonanni B, Gandini S. Metformin and cancer risk in diabetic patients: a systematic review and meta-analysis. Cancer Prev Res (Phila). 2010 Nov;3(11):1451-61. doi: 10.1158/1940-6207.CAPR-10-0157. Epub 2010 Oct 12. PMID 20947488
- [Background] Jiralerspong S, Palla SL, Giordano SH, Meric-Bernstam F, Liedtke C, Barnett CM, Hsu L, Hung MC, Hortobagyi GN, Gonzalez-Angulo AM. Metformin and pathologic complete responses to neoadjuvant chemotherapy in diabetic patients with breast cancer. J Clin Oncol. 2009 Jul 10;27(20):3297-302. doi: 10.1200/JCO.2009.19.6410. Epub 2009 Jun 1. PMID 19487376
- [Background] Towler MC, Hardie DG. AMP-activated protein kinase in metabolic control and insulin signaling. Circ Res. 2007 Feb 16;100(3):328-41. doi: 10.1161/01.RES.0000256090.42690.05. PMID 17307971
- [Background] Vazquez-Martin A, Oliveras-Ferraros C, del Barco S, Martin-Castillo B, Menendez JA. mTOR inhibitors and the anti-diabetic biguanide metformin: new insights into the molecular management of breast cancer resistance to the HER2 tyrosine kinase inhibitor lapatinib (Tykerb). Clin Transl Oncol. 2009 Jul;11(7):455-9. doi: 10.1007/s12094-009-0384-0. PMID 19574203
- [Background] Vazquez-Martin A, Oliveras-Ferraros C, Lopez-Bonet E, Menendez JA. AMPK: Evidence for an energy-sensing cytokinetic tumor suppressor. Cell Cycle. 2009 Nov 15;8(22):3679-83. doi: 10.4161/cc.8.22.9905. Epub 2009 Nov 24. PMID 19844168
- [Background] O'Toole D, Ducreux M, Bommelaer G, Wemeau JL, Bouche O, Catus F, Blumberg J, Ruszniewski P. Treatment of carcinoid syndrome: a prospective crossover evaluation of lanreotide versus octreotide in terms of efficacy, patient acceptability, and tolerance. Cancer. 2000 Feb 15;88(4):770-6. doi: 10.1002/(sici)1097-0142(20000215)88:43.0.co;2-0. PMID 10679645
- [Background] CLARINET Abstract E17-7103, Amsterdam EJC, vol 49 (3), 2013
- [Background] Martin-Richard M, Massuti B, Pineda E, Alonso V, Marmol M, Castellano D, Fonseca E, Galan A, Llanos M, Sala MA, Pericay C, Rivera F, Sastre J, Segura A, Quindos M, Maisonobe P; TTD (Tumores del Tracto Digestivo) Study Group. Antiproliferative effects of lanreotide autogel in patients with progressive, well-differentiated neuroendocrine tumours: a Spanish, multicentre, open-label, single arm phase II study. BMC Cancer. 2013 Sep 20;13:427. doi: 10.1186/1471-2407-13-427. PMID 24053191
- [Background] Machin, D., Campbell, M., Fayers, P., and Pinol, A. 1997. Sample Size Tables for Clinical Studies, 2nd edition. Blackwell Science. Malden, MA.
- [Background] Cohen J. (1988) Statistical Power Analysis fo the Behavioural Sciences, Lawrence Erbaum Associates, Hillsdale, New Jersey.
- [Background] NCSS (Number Cruncher Statistical System) Versione 8.0.2012.
- [Background] Hintze, J. (2011). PASS (Power Analysis and Sample Size System) 11. NCSS, LLC. Kaysville, Utah, USA.
- [Background] Chow, S.C.; Shao, J.; Wang, H. 2003. Sample Size Calculations in Clinical Research. Marcel Dekker. New York
- [Background] Fleiss, J. L., Levin, B., Paik, M.C. 2003. Statistical Methods for Rates and Proportions. Third Edition. John Wiley & Sons. New York.
- [Background] Lachin, John M. 2000. Biostatistical Methods. John Wiley & Sons. New York.
- [Background] - Zar, Jerrold H. 1984. Biostatistical Analysis (Second Edition). Prentice-Hall. Englewood Cliffs, New Jersey
- [Background] Shackelford DB, Shaw RJ. The LKB1-AMPK pathway: metabolism and growth control in tumour suppression. Nat Rev Cancer. 2009 Aug;9(8):563-75. doi: 10.1038/nrc2676. PMID 19629071
- [Background] Lippitz BE. Cytokine patterns in patients with cancer: a systematic review. Lancet Oncol. 2013 May;14(6):e218-28. doi: 10.1016/S1470-2045(12)70582-X. PMID 23639322
- [Background] Korsse SE, Peppelenbosch MP, van Veelen W. Targeting LKB1 signaling in cancer. Biochim Biophys Acta. 2013 Apr;1835(2):194-210. doi: 10.1016/j.bbcan.2012.12.006. Epub 2012 Dec 31. PMID 23287572
- [Background] Lin CC, Yeh HH, Huang WL, Yan JJ, Lai WW, Su WP, Chen HH, Su WC. Metformin enhances cisplatin cytotoxicity by suppressing signal transducer and activator of transcription-3 activity independently of the liver kinase B1-AMP-activated protein kinase pathway. Am J Respir Cell Mol Biol. 2013 Aug;49(2):241-50. doi: 10.1165/rcmb.2012-0244OC. PMID 23526220
- [Background] Vlotides G et al. "In Vitro Anticancer Effect of Metformin in Neuroendocrine Tumour Cells" Abstract B9; 10th Annual ENETS Conference, 6-8 March 2013, Barcelona
- [Background] Marciello F. et al. "Role of Metformin on Recurrence-Free-Survival (RFS) in Neuroendocrine Tumors (NETs)" Abstract M4; 11th Annual ENETS Conference, 5-7 March 2014, Barcelona
- [Background] S. Pusceddu, et al. "Metformin impact on progression-free survival in advanced pancreatic well-differentiated neuroendocrine tumors (pWDNETs). Retrospective evaluation in diabetic patients receiving Everolimus plus Octreotide LAR treatment" 1146Tip - 39th ESMO Congress, Madrid - Annals of Oncology, Vol 25, Suppl 4, 2014
- [Background] F.G.M. De Braud, et al. "Activity and safety of Everolimus in combination with Octreotide LAR and Metformin in patients with advanced pancreatic well-differentiated Neuroendocrine Tumors (pWDNETs): a single-center, open-label, phase II, proof-of-concept study (MetNET1 trial)"; 1163Tip - 39th ESMO Congress, Madrid - Annals of Oncology, Vol 25, Suppl 4, 2014
- [Background] Custodio A et al. "Prognostic Role of Diabetes Mellitus (DM) and Metformin (MET) Therapy in Patients (pts) with Advanced G1-G2 Neuroendocrine Tumors (NETs) Treated with Everolimus (EVE)" - abstract L7, ENETS 2015
- [Background] Custodio A et al. "Everolimus (EVE)-Induced Hyperglycemia (HG) in Patients (pts) with Advanced G1-G2 Neuroendocrine Tumors (NETs): Clinical Relevance and Predictive Value" - abstract L8, ENETS 2015
- [Background] Colao AM et al. "Metformin-Based Oral Antidiabetic Therapy Is Effective at Controlling Hyperglycemia Associated with Pasireotide in Patients with Acromegaly" - abstract PP09-2 - ENDO 2015
- [Background] Colao A, Auriemma RS, Savastano S, Galdiero M, Grasso LF, Lombardi G, Pivonello R. Glucose tolerance and somatostatin analog treatment in acromegaly: a 12-month study. J Clin Endocrinol Metab. 2009 Aug;94(8):2907-14. doi: 10.1210/jc.2008-2627. Epub 2009 Jun 2. PMID 19491229
- [Background] Rodbard HW, Blonde L, Braithwaite SS, Brett EM, Cobin RH, Handelsman Y, Hellman R, Jellinger PS, Jovanovic LG, Levy P, Mechanick JI, Zangeneh F; AACE Diabetes Mellitus Clinical Practice Guidelines Task Force. American Association of Clinical Endocrinologists medical guidelines for clinical practice for the management of diabetes mellitus. Endocr Pract. 2007 May-Jun;13 Suppl 1:1-68. doi: 10.4158/EP.13.S1.1. No abstract available. PMID 17613449
- [Background] Einhorn D, Reaven GM, Cobin RH, Ford E, Ganda OP, Handelsman Y, Hellman R, Jellinger PS, Kendall D, Krauss RM, Neufeld ND, Petak SM, Rodbard HW, Seibel JA, Smith DA, Wilson PW. American College of Endocrinology position statement on the insulin resistance syndrome. Endocr Pract. 2003 May-Jun;9(3):237-52. No abstract available. PMID 12924350
- [Background] Modlin IM, Pavel M, Kidd M, Gustafsson BI. Review article: somatostatin analogues in the treatment of gastroenteropancreatic neuroendocrine (carcinoid) tumours. Aliment Pharmacol Ther. 2010 Jan 15;31(2):169-88. doi: 10.1111/j.1365-2036.2009.04174.x. Epub 2009 Oct 21. PMID 19845567
- [Result] Jiao Y, Shi C, Edil BH, de Wilde RF, Klimstra DS, Maitra A, Schulick RD, Tang LH, Wolfgang CL, Choti MA, Velculescu VE, Diaz LA Jr, Vogelstein B, Kinzler KW, Hruban RH, Papadopoulos N. DAXX/ATRX, MEN1, and mTOR pathway genes are frequently altered in pancreatic neuroendocrine tumors. Science. 2011 Mar 4;331(6021):1199-203. doi: 10.1126/science.1200609. Epub 2011 Jan 20. PMID 21252315
- [Result] Wolin EM. The expanding role of somatostatin analogs in the management of neuroendocrine tumors. Gastrointest Cancer Res. 2012 Sep;5(5):161-8. PMID 23112884